CLINICAL TRIAL: NCT02359162
Title: Comparison of Gemcitabine, Oxaliplatin and Pegaspargase and Etoposide, Vincristine, Doxorubicin, Cyclophosphamide and Prednisone as First-line Chemotherapy in Patients With NK/T-cell Lymphoma：a Prospective Randomized Phase III Study
Brief Title: Efficacy and Safety Study of P-Gemox vs.EPOCH as First-line Chemotherapy to Treat NK/T-cell Lymphoma With Early Stage
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is out of date
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wanghua, Professor of departments of Department of Hematological Oncology, Sun Yat-sen University Cancer Center., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-NK-308
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
Keywords: NK/T-cell lymphoma; induction chemotherapy; survival
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gemcitabine; Oxaliplatin; pegaspargase; Etoposide; Vincristine; Doxorubicin; Cyclophosphamide; Prednisone; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P-Gemox (Experimental): P-Gemox:gemcitabine :1250mg/m2 (ivdrip) on days 1, oxaliplatin :85 mg/m2 (ivdrip) on day 1, and pegaspargase : 2500 IU/m2 (intramuscular injection) on day 1.Cycle is repeated every 14 days.
  IMRT：IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50 grays (Gy) in 25 fractions.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Pegaspargase; Radiation: IMRT
- EPOCH (Active Comparator): EPOCH:Patients received the EPOCH chemotherapy regimen every 3 weeks. The EPOCH regimen included a 24 h continuous infusion of etoposide (50 mg/m 2 /day), vincristine (0.4 mg/m 2 /day) and doxorubicin(10 mg/m 2 /day administered on days 1-4, followed by cyclophosphamide (750 mg/m2 /day) over 15 min intravenously on day 5 and prednisone (60 mg/m 2 /day) on days1- 5 orally.
  IMRT：IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50 grays (Gy) in 25 fractions.
  Interventions: Drug: Etoposide; Drug: Vincristine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Prednisone; Radiation: IMRT

INTERVENTIONS:
Drug: Gemcitabine — gemcitabine :1250mg/m2 (ivdrip) on days 1
  Arms: P-Gemox
Drug: Oxaliplatin — oxaliplatin :85 mg/m2 (ivdrip) on day 1
  Arms: P-Gemox
Drug: Pegaspargase — pegaspargase : 2500 IU/m2 (intramuscular injection)
  Arms: P-Gemox
Drug: Etoposide — 50 mg/m 2 /day 24 h continuous infusion on days 1-4
  Arms: EPOCH
Drug: Vincristine — 0.4 mg/m 2 /day 24 h continuous infusion on days 1-4
  Arms: EPOCH
Drug: Doxorubicin — 10 mg/m 2 /day 24 h continuous infusion on days 1-4
  Arms: EPOCH
Drug: Cyclophosphamide — cyclophosphamide 750 mg/m2 /day over 15 min intravenously on day 5
  Arms: EPOCH
Drug: Prednisone — 60 mg/m 2 /day 60 mg/m 2 /day on days 1-5
  Arms: EPOCH
Radiation: IMRT — IMRT is delivered using 6-8 MeV linear accelerator using intensity-modulated radiation treatment planning. The radiation dose is 50 grays (Gy) in 25 fractions.
  Other Names: Intensity-modulated radiation therapy

SUMMARY:
Purpose :To compare the efficacy and and safety of the P-Gemox chemotherapy regimen with those of the EPOCH regimen for stage IE to IIE ENKTL.

DETAILED DESCRIPTION:
ENKTL is an aggressive type of NHL characterized by poor survival, for which the optimal treatment strategies have not been fully defined. Radiation therapy (RT) is widely administered for patients with localized nasal disease, and produces a complete response (CR) rate of up to 70%.However, local and systemic failures are observed frequently in patients who receive RT alone.Therefore, chemotherapy is needed in combination with RT to reduce the risk of recurrence. Unfortunately, ENKTL shows a poor response to the CHOP chemotherapy regimen (cyclophosphamide, doxorubicin, vincristine and prednisone) . EPOCH (etoposide, vincristine, doxorubicin, cyclophosphamide and prednisone) chemotherapy followed by involved field radiotherapy (IFRT) results in a CR rate of 75.0%. Recently, a chemotherapy regimen including gemcitabine,oxaliplatin and l-asparaginase (GELOX) has emerged, with promising results.Since 2003, a proportion of patients newly diagnosed with ENKTL were treated with the EPOCH chemotherapy regimen at some hospitals in China. From 2008, many hospitals in the southern part of China began to use the GELOX( Pegaspargase is used instead of l-asparaginase,P-Gemox).Our multicenter retrospective study showed the GELOX regimen produces a better long outcome with less toxicity than the EPOCH regimen for patients with early stage ENKTL.However,further prospective randomized clinical trials are needed to confirm the conclusion.

1. Patients

   * All patients should sign a written informed consent form before enrollment, and the study should be approved by the Sun Yat-sen University Cancer Center Ethics Board.
   * Baseline of patients: Computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, and bilateral bone marrow aspiration or biopsy. Positron emission tomography-CT scans (optional). Epstein-Barr virus (E B V) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA), β2-micro globulin (β2-MG) , IL-9 and IL-15 in the serum.
   * Recheck before and after every course: Epstein-Barr virus (EBV) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA), β2-micro globulin (β2-MG), IL-9 and IL-15 in the serum.
   * Recheck every two course: Computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, and bilateral bone marrow aspiration or biopsy. Positron emission tomography-CT scans (optional)
2. Treatment Protocol:

   * The GELOX regimen consist of the following drugs: gemcitabine ：1250 mg/ m2 on days 1,ivdrip oxaliplatin ：85 mg/m2 on day 1, ivdrip pegaspargase : 2500 IU/m 2 daily on day 1,intramuscular. The treatment cycle is repeated every 14 days.
   * The EPOCH regimen included a 24 h continuous infusion of etoposide (50 mg/m 2 /day), vincristine (0.4 mg/m 2 /day) and doxorubicin(10 mg/m 2 /day administered on days 1-4, followed by cyclophosphamide (750 mg/m2 /day) over 15 min intravenously on day 5 and prednisone (60 mg/m 2 /day) 60 mg/m 2 /day on days 1-5.The treatment cycle is repeated every 21 days.

After at least two cycles of chemotherapy, patients who have achieved stable disease (SD) following two cycles, partial response (PR) after four cycles or complete response (CR) after six cycles of chemotherapy are referred to primary IFRT.

◦IFRT was delivered using 6-MeV linear accelerator using 3-dimensional conformable treatment planning. The IFRT dose was 56 grays (Gy) in 28 fractions, we define the clinical target volume of limited stage IE disease as the bilateral nasal cavity, bilateral ethmoid sinuses, and ipsilateral maxillary sinus; and the clinical target volume would extend to involved tissues for patients who had extensive stage IE disease. For patients who had stage IIE disease, the clinical target volume also, included the bilateral cervical lymph node area.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-69years
* Ann Arbor stage IE,or stage IIE with cervical lymph node involvement
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.
* primary lesion not from the upper respiratory

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)
  time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first

SECONDARY OUTCOMES:
complete remission rate | every 4 weeks,up to completion of treatment(approximately 6 months)
  The criteria for the efficacy evaluation (overall response rate and complete remission) of the regimen is according to the following article:
  Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999;17:1244.
overall survival | .up to end of follow-up-phase (approximately 3 years)
  overall survival (OS): time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first
safety, as measured by adverse events | up to end of follow-up-phase (approximately 3 years)
  including hematological safety and non-hematological safety.All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

OTHER OUTCOMES:
serum Epstein-Barr virus(EBV) DNA copies | every 3 weeks,up to completion of treatment(approximately 6 months)
serum β2-microglobulin | every 3 weeks,up to completion of treatment(approximately 6 months)
serum interleukin 9 | every 3 weeks,up to completion of treatment(approximately 6 months)
serum interleukin 15 | every 3 weeks,up to completion of treatment(approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD., Principal Investigator — Department of Hematological Oncology, Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Wang H, Wuxiao ZJ, Zhu J, Wang Z, Wang KF, Li S, Chen X, Lu Y, Xia ZJ. Comparison of gemcitabine, oxaliplatin and L-asparaginase and etoposide, vincristine, doxorubicin, cyclophosphamide and prednisone as first-line chemotherapy in patients with stage IE to IIE extranodal natural killer/T-cell lymphoma: a multicenter retrospective study. Leuk Lymphoma. 2015 Apr;56(4):971-7. doi: 10.3109/10428194.2014.939964. Epub 2014 Aug 20. PMID 24991715
- [Result] Wang L, Wang ZH, Chen XQ, Li YJ, Wang KF, Xia YF, Xia ZJ. First-line combination of gemcitabine, oxaliplatin, and L-asparaginase (GELOX) followed by involved-field radiation therapy for patients with stage IE/IIE extranodal natural killer/T-cell lymphoma. Cancer. 2013 Jan 15;119(2):348-55. doi: 10.1002/cncr.27752. Epub 2012 Jul 18. PMID 22811078
- [Result] Huang H, Lin Z, Lin X, Cai Q, Xia Z, Jiang W. Long-term outcomes of patients with newly diagnosed extranodal natural killer/T-cell lymphoma treated by etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin regimen: a single-institution experience. Leuk Lymphoma. 2011 Jun;52(6):1041-8. doi: 10.3109/10428194.2011.561388. PMID 21599590
- See also: medlineplus — http://www.nlm.nih.gov/medlineplus/
- See also: drug imformation — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp